CLINICAL TRIAL: NCT06258408
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Profiles and Efficacy of Oral BB102 Tablets in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of BB102 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Broadenbio Ltd., Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB102-ST-Ⅰ-02
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
Keywords: BB102; FGFR4; First-in-Human; Dose Escalation; FGF19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BB102 monotherapy (Experimental): The study is composed of fasted dose cohorts and fed dose cohort. BB102 will be administered orally daily alone as monotherapy in all cohorts. In the fasted dose cohorts, the subjects will receive once daily of BB102 monotherapy fasted across approximately 6 ascending dose levels. The starting dose is 50mg/day. In the fed dose cohort, the subjects will receive once daily of BB102 monotherapy in a fed condition. The dose selected for fed dose cohort must be deemed safe as assessed by safety monitoring committee (SMC).
  Interventions: Drug: BB102 tablet

INTERVENTIONS:
Drug: BB102 tablet — BB102 tablets will be administered orally once daily(QD).
  Other Names: BB102

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, efficacy and preliminary food effect of BB102, a highly selective and potent FGFR4 inhibitor, as monotherapy in subjects with advanced solid tumors. This study has two phase: dose escalation phase and expansion phase.

DETAILED DESCRIPTION:
This first-in-human (FIH) study of BB102 will evaluate safety, tolerability, pharmacokinetics (PK), efficacy and preliminary food effect in subjects with advanced solid tumors. In dose escalation trial, the primary objective is to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of BB102 as monotherapy, and to evaluate the safety and tolerability of BB102. The secondary objectives include the assessments of PK profile, preliminary efficacy, preliminary food effect (FE), preliminary metabolites identification, biomarkers and C-QTcF analysis of BB102. In expansion trial, the primary objective is to evaluate the efficacy of BB102 in subjects with FGF19 or FGFR4 positive advanced primary hepatocellular carcinoma (HCC) or other advanced solid tumors. The secondary objectives include the assessments of PK profile, safety and biomarkers of BB102.

ELIGIBILITY:
Inclusion Criteria:

1. For the dose escalation trial, histologically, cytologically confirmed or clinically confirmed advanced solid tumors patients who without available standard treatment, have disease progression on standard treatment or cannot tolerate standard treatment.

   For the expansion trial, histologically or cytologically confirmed FGF19 or FGFR4 positive advanced primary HCC or other advanced solid tumors patients who without available standard treatment, have disease progression on standard treatment or cannot tolerate standard treatment.
2. For the dose escalation trial, at least one evaluable lesion as defined by RECIST v1.1.

   For the expansion trial, at least one measurable lesion as defined by RECIST v1.1.
3. Eastern Cooperative Oncology Group (ECOG) score ≤1.
4. Expected survival ≥ 3 months.
5. Adequate organ function.
6. Female subjects of childbearing potential must have a negative pregnancy test prior to the first dose and are required to use effective contraception from signing the ICF until 6 months after the last dose of study treatment.
7. Fully informed of the study and voluntarily signed the informed consent form (ICF), and willing to follow and have the ability to complete all trial procedures.

Exclusion Criteria:

1. Use of systemic immunosuppressive or systemic cortisol (≥10 mg prednisone or other equivalent hormones) within 4 weeks.
2. Prior use of selective FGFR4 inhibitor and/or pan-FGFR inhibitor therapy.
3. Use of cytotoxic chemotherapeutics within 4 weeks, OR use of state-approved Chinese traditional patent drugs/Chinese traditional drugs with an antitumor effect within 2 weeks.
4. Anti-tumor endocrine therapy, radiotherapy, interventional embolization, radiofrequency, proton therapy, radioimmunotherapy, immunotherapy or other biotherapies within 4 weeks.
5. Use of other clinical investigational drug or therapy that was not marketed within 4 weeks.
6. The patient is receiving drugs or therapies prohibited in the protocol and cannot discontinue such use at least 2 weeks.
7. Pregnant or lactating females.
8. Presence of clinically significant gastrointestinal disorder that may affect the intake, transport, or absorption of the study drug at screening.
9. Patient with dual-source cancer within 5 years.
10. Presence of clinically symptomatic metastases to the central nervous system or meninges or other evidence showing that metastatic lesions in the central nervous system or meninges have not yet been controlled at screening, which, at the investigator's discretion, is not suitable for enrollment.
11. History of severe neurological or psychiatric disorders, including epilepsy, dementia, moderate to severe depression, etc.
12. Clinically significant and uncontrolled cardiovascular diseases.
13. Pulmonary embolism within 6 months.
14. Prior allogeneic stem cell transplantation, bone marrow transplantation or vital organ transplantation.
15. Presence of uncontrollable infectious disease, congenital immunodeficiency disease,acquired immunodeficiency syndrome, syphilis, active hepatitis B, hepatitis C virus (HCV) infection.
16. Severe active infection, including but not limited to bacteremia, severe pneumonia, etc., occurred within 2 weeks; an active infection that received therapeutic intravenous antibiotics within 2 weeks.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | Single dose to the end of Cycle 1 (each cycle is 21 days)
  To assess the safety and tolerability of BB102 tablet as monotherapy in subjects with advanced solid tumors and to determine the maximum tolerated dose (MTD) of BB102 tablet, and to provide a basis for determination of the recommended dose (RP2D) for Phase II clinical trials.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28 to Day -1) through up to 12 months or until disease progression
  AEs and SAEs will be characterized by type, seriousness, relationship to study treatment, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) and timing.
  FGF19 or FGFR4 positive advanced primary HCC or other advanced solid tumors.

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: Peak Plasma Concentration (Cmax) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Time to Peak Concentration (Tmax) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Area under the plasma concentration-time curve (AUC) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Elimination half-life (t½) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Objective response rate (ORR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Duration of response (DOR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Disease control rate (DCR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Progression-free survival (PFS) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, MD, Principal Investigator — Henan Cancer Hospital
Locations (2):
- China (2):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan

DOCUMENTS (2):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT06258408/Prot_000.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT06258408/ICF_001.pdf